CLINICAL TRIAL: NCT01791452
Title: Novel Association of Cholesterol Ester Storage Disease Due to Lysosomal Acid Lipase Deficiency and Non-Alcoholic Fatty Liver Disease: A Prospective Clinical Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assy Nimer (Other Government)
Responsible Party: Sponsor-Investigator, Assy Nimer, MD, Ziv Hospital
Organization: Ziv Hospital (Other Government)
Other Study IDs: 0042-12-ZIV
Record Dates: First submitted 2013-02-10; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Non-alcoholic Fatty Liver Disease; Cholesterol Ester Storage Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Cholesterol Ester Storage Disease

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- NAFLD

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a world-wide problem with a global prevalence estimated at 1.5 billion people. It is characterised by significant diversity and phenotypic heterogeneity. Morbidity rates are estimated at 20% to 30% in Western adults, increasing to 90% in patients who are morbidly obese or diabetic. Risk factors in non-obese NAFLD patients are of especial practical and theoretical importance. Cholesterol Ester Storage Disease (CESD) is an autosomal recessive chronic disease of variable phenotype, caused by a deficiency in lysosomal acid lipase (LAL) and characterized by accumulation of fat in tissues and organs. Hepatic accumulation of fat in this disorder can cause hepatomegaly with varying degrees of damage varying from steatosis to fibrosis, elevated aminotransaminases, and isolated splenomegaly. Since the contribution of LAL deficiency to non-obese NAFLD is poorly understood, the investigators propose to evaluating the association between NAFLD and LAL deficiency in a prospective study in our population.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80 years;
* BMI 25-40;
* Fatty liver disease (bright liver, hepatomegaly by ultrasound (Liver span > 15 cm mid clavicle line), splenomegaly (>13 cm) or both.

Exclusion Criteria:

* Alcohol abuse>30 gm/day, or > 70 gram per week;
* Soft drink abuse;
* Drugs known to cause fatty liver;
* Chronic hepatitis (B and C);
* Biliary liver disease;
* Autoimmune hepatitis;
* HIV;
* Genetic/Metabolic liver disease (Wilson, alpha-1 antitrypsin, CF);
* Failure to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 subjects will be enrolled and informed consent obtained. After clinical evaluation, subjects will undergo liver ultrasound, non-invasive liver elastography (Fibroscan) and standard biochemical evaluation including glucose, insulin, TG, HDL, LDL, leptin, adiponectin and TNF-alpha. They will then be divided into 2 groups: NAFLD, and NAFLD with fibrosis (NASH). In addition a cohort of healthy volunteers will also be studied. LAL activity in dry blood spots (DBS) will be measured using the substrate 4-methylumbelliferyl palmitate. LAL activity will be measured by measuring total lipase activity and lipase activity in the presence of Lalistat2.
Sampling Method: Probability Sample
Dates: Primary Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
liver ultrasound, ultrasound Doppler of the common carotid artery, hepatic Fibroscan evaluation (transient elastography) for assessment of steatosis and fibrosis | year

CONTACTS AND LOCATIONS:
Locations (1):
- Assy Nimer, Safed, Israel, Israel